CLINICAL TRIAL: NCT04756206
Title: Role of Dutasteride in Treatment of Category IIIB Chronic Prostatitis (A Placebo-Controlled Study)
Brief Title: Role of Dutasteride in Treatment of Chronic Prostatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21/2020
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Dutasteride; Category IIIB Chronic Prostatitis
MeSH Terms: interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dutasteride (Active Comparator): Dutasteride of 0.5 mg once daily was given for 3 months compared to a placebo.
  Interventions: Drug: Dutasteride 0.5 mg
- Placebo (Placebo Comparator): same form and color of Dutasteride tablet was given at the same regimen to act as a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride 0.5 mg — patients were randomized into 2 equal groups with 1:1 ratio using a computer-based system. Dutasteride of 0.5 mg once daily was given for 3 months compared to a placebo. Patients, data collector,s and the statistician were blinded to the type of intervention.
  Arms: Dutasteride
Drug: Placebo — patients were randomized into 2 equal groups with 1:1 ratio using a computer-based system. Dutasteride of 0.5 mg once daily was given for 3 months compared to a placebo. Patients, data collector,s and the statistician were blinded to the type of intervention.
  Arms: Placebo

SUMMARY:
this placebo controlled study aims to evaluate the efficacy of Dutasteride in the management of Chronic prostatitis type 3.

DETAILED DESCRIPTION:
Nonbacterial prostatitis refers to a condition that affects patients who present with symptoms of prostatitis without a positive culture for urine or expressed prostate secretions (EPS). With time our understanding of prostatitis was evolved to include a different clinical phenotype with a variety of voiding presentation and symptomatology rather than just inflammation and infection. The two main clinical presentations of prostatitis include pelvic pain and LUTS.

The National Institutes of Health and the National Institute of Diabetes and Digestive and Kidney Diseases (NIH-NIDDK) proposed the first classification of prostatitis into 4 categories in 1995 that was later published in 1998. Bacterial prostatitis represented category I and III while nonbacterial prostatitis including chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) was categorized as category III that was further subdivided into class IIIa (inflammatory CPPS) and b (non-inflammatory CPPS). Category IV encompasses asymptomatic inflammatory prostatitis.

Shoskes et al, mentioned that inflammation and the upregulation of cytokine expression and release in the prostate secondary to an inflammatory process led to the presenting symptoms in such a condition. The recently introduced UPOINT phenotype categorization of CP/CPPS (Urinary, Psychosocial, Organ-specific, Infection, Neurological/Systemic, Tenderness of the skeletal muscles). This categorization shows up to 60% of men have at least prostate organ associated symptoms.

The prostate lies under the hormonal control of dihydrotestosterone (DHT); thus 5 alpha-reductase inhibitors (5ARIs) might be beneficial in the treatment of prostatitis. Dutasteride is a 5α-reductase inhibitor, and hence is a type of anti-androgen. It works by decreasing the production of (DHT) in certain parts of the body like the prostate gland. It inhibits all three forms of 5α-reductase and can decrease DHT levels in the blood by up to 98%.

5ARIs have been previously evaluated on a narrow scale in the management of prostatitis with promising results of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 40 and 70 years old, diagnosed with chronic prostatitis based on the presence of pelvic pain for ≥3 months of the preceding 6 months

Exclusion Criteria:

Patients with bacterial prostatitis

* documented site of infection along the urinary tract,
* urinary bladder tumors
* prostate cancer
* previous history of pelvic radiation or chemotherapy were excluded from our study.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Chronic prostatitis is a disease that affects men only.
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
NIH chronic prostatitis symptom index in study population | assessment was made before treatment
  scoring system aims to evaluate chronic prostatitis and severity of symptoms
NIH chronic prostatitis symptom index in study population | assessment was made at 3 months after intervention
  scoring system aims to evaluate chronic prostatitis and severity of symptoms

SECONDARY OUTCOMES:
change in libido in study population | 3 months after medication
  according to sexual desire inventory -2
Gastritis in study population | 3 months after medication
  side effect of medication (if present or not)
Dizziness in study population | 3 months after medication
  side effect of medication (if present or not)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Higazy A, Shorbagy AA, Shabayek M, Radwan A, Halim GN, Osman D, Osman T. Short course of dutasteride in treatment of a refractory category IIIB chronic prostatitis (A placebo-controlled study). Prostate Int. 2022 Dec;10(4):213-217. doi: 10.1016/j.prnil.2022.06.002. Epub 2022 Jun 20. PMID 36570649